CLINICAL TRIAL: NCT05997277
Title: A Pilot Study Evaluating the Safety and Efficacy of Deucravacitinib Compared to Placebo in the Treatment of Moderate-to-severe Hidradenitis Suppurativa (HS).
Brief Title: Evaluating the Safety and Efficacy of Deucravacitinib Compared to Placebo Hidradenitis Suppurativa (HS).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn by sponsor due to funding priorities, study cannot continue without funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Alexa B Kimball, Professor of Dermatology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P000400
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deucravacitinib - Study Drug (Experimental): Deucravacitinib group: 6 mg po bid x 16 weeks
  Interventions: Drug: Deucravacitinib
- Placebo (Placebo Comparator): Placebo group: 1 tablet po bid x 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Deucravacitinib is a stable deuterium-containing compound (where deuterium is a stable, nonradioactive isotope of hydrogen) and a potent, highly selective small molecule inhibitor of TYK2. Deucravacitinib has a unique mode of binding that provides the high selectivity over the other members of the JAK family of nonreceptor tyrosine kinases. 1 active oral tablet (6mg) in the morning and evening for 16weeks.
  Other Names: BMS-986165; SOTYKTU
  Arms: Deucravacitinib - Study Drug
Drug: Placebo — Placebo will consist of a tablet (0mg) and will be administered orally BID for 16weeks.
  Arms: Placebo

SUMMARY:
The study is a randomized, proof of concept study. 30 patients aged 18 and over with HS will be included in this single center, randomized, double-blind, parallel-group study. Dosage of deucravacitinib will be given according to the investigational regimen as follows: 6 mg po bid for 16 weeks. The study compromises a 4-week screening period, a 16-week study period, and a 4-week follow-up period. The follow-up period consists of a follow-up phone call 4 weeks after the last study drug dose.

DETAILED DESCRIPTION:
The objective of this study is to investigate the efficacy of Deucravacitinib (BMS- 986165) in the treatment of Hidradenitis Suppurativa.

Subjects will be randomly assigned to receive either Deucravacitinib (6 mg twice daily) or placebo for 16 weeks. Assessments will be performed at Baseline and weeks 4, 8, 12, and 16 by a blinded investigator. During this visits, subjects will also be asked to complete a quality of life questionnaire (DLQI) and Visual Analog Scale (VAS) for pain.

A total enrollment of 30 subjects (20 study drug, 10 placebo) is anticipated in this single- center, randomized, double-blind, parallel-group study. This study powered to show a significant difference in efficacy of treatment using the following assumptions based on other clinical trials: baseline average inflammatory lesion count of 12, improvement of 7 in the treatment group and 3 in the placebo group, with a power of 0.87, SD of 3.25 and alpha level of 0.05. The HiSCR will be a secondary endpoint (reduction of inflammatory lesions by 50% with no increase in fistulas or abscesses).

ELIGIBILITY:
Inclusion Criteria:

* • Male or Female at least 18 -70 years of age

  * Able to provide informed consent
  * Have at least 5 abscesses and/or inflammatory nodule (AN) count at baseline visits
  * Have HS lesions in 2 distinct anatomical areas
  * Women of Childbearing potential must have a negative serum urine pregnancy test at screening and a negative urine pregnancy test at baseline -- prior to administration of the first dose of study medication
  * Women of childbearing potential must be willing to continue a highly effective method of birth control throughout the study (oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal foam/gel/film/cream/suppository (if available in their locale); male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence (when this is in line with the preferred and usual lifestyle of the participant).
  * Tuberculosis Screening

    * Negative IGRA screening for tuberculosis within 3 months prior to screening, OR
    * If a positive history of latent tuberculosis:
* Currently receiving treatment for latent TB per standard of care (with at least 4 weeks of treatment prior to baseline visit)
* Have documentation of having completed treatment within 5 years prior to baseline • Agree not to have a live vaccination during the study

Exclusion Criteria:

* • Any other active skin disease that in the opinion of the investigator would interfere with the assessment of HS

  * Have greater than 20 draining fistula at baseline
  * Receipt of non-biologic treatments for HS within 4 weeks prior to baseline other than antibiotics or hormonal therapy
  * Receipt of TNF agents (i.e. Infliximab, adalimumab) or other biologics within 6 weeks prior to baseline
  * Receipt of new hormonal therapy for HS within 3 weeks prior to baseline
  * Receipt of oral antibiotics within 3 weeks prior to baseline.

    o NOTE: subjects on concomitant antibiotics with a stable dose for 4 weeks prior to baseline visit may be included in the study. Only 25% of total enrollment may be on concomitant antibiotics.
  * Receipt of intralesional kenalog injections within 2 weeks prior to baseline
  * Receipt of topical steroids or topical antibiotics for HS for 2 weeks prior to baseline

    o NOTE: subjects may continue topical washes (benzoyl peroxide, chlorhexidine, zinc pyrithione, dilute bleach)
  * Receipt of opioid analgesics or other concomitant analgesics for HS pain within 72 hours prior to the baseline visit

    o Concomitant use of non-opioid analgesics for treatment of chronic non-HS pain is allowed as long as the dose has been stable for 14 days prior to baseline and expected to remain constant throughout the study
  * Any uncontrolled diagnosis or condition that in the opinion of the investigator will interfere with the assessments or the study.
  * Currently has a malignancy or a history of a malignancy within 5 years before screen (except successfully treated non-melanoma skin cancer or cervical carcinoma in situ)
  * History of an ongoing, chronic or recurrent infectious disease
  * Are currently pregnant, breastfeeding, or planning to get pregnant during the study

    o male participants who are actively trying to conceive with their partner are also excluded.
  * Previous hypersensitivity reaction to deucravacitinib or to any of the components
  * Known allergy to tetracycline antibiotics
  * Known infection with HIV, hepatitis B or hepatitis C at screening or randomization. Patients who are Hepatitis B Core antibody and/or Hep B Surface Antigen positive will be excluded from this study. Patients who are Hepatitis C ab positive will also be excluded from this study.
  * Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Inflammatory lesion counts (including combined counts of inflammatory nodules (N) and abscesses (A)/AN count) at week 16. | Baseline and Week 16
  We will assess the average change in inflammatory lesion count per subject following 16 weeks of treatment as compared to baseline. Inflammatory lesions are defined as inflammatory nodules or abscesses.

SECONDARY OUTCOMES:
The population treatment effect on proportion of participants with Hidradenitis Suppurativa Clinical Response (HiSCR) at week 16 for the active treatment group relative to placebo without regard to IP compliance | Baseline and Week 16
  The number and proportion of participants who achieve a HiSCR at Weeks 16 will be summarized and compared to placebo. HiSCR is a validated, binary outcome and is defined as at least a 50% reduction from baseline in the total abscess and inflammatory- nodule count, with no increase in the abscess or draining fistula count.
  HiSCR Assessment Relative to baseline, all three criteria must be met.
  1. >50% reduction in the total number of inflammatory nodules and abscesses
  2. No increase in abscess count
  3. No increase in draining fistula count
Changes in IHS4 scores at weeks 4, 8, 12, and 16 compared to baseline. | Baseline, weeks 4, 8, 12, and 16
  The novel IHS4 is a validated tool to dynamically assess HS severity and can be used both in real-life and the clinical trials setting.
  The resulting IHS4 score is arrived at by the number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild, 4-10 signifies moderate and 11 or higher signifies severe disease.
Changes in Hurley Stage scores at weeks 4, 8, 12, and 16 compared to baseline. | Baseline, weeks 4, 8, 12, and 16
  Hurley Staging is a surgical staging system used to describe disease severity. No improvement in Hurley scoring is expected with medical management alone. Pre- and post-study drug scores will be compared.
  The Hurley clinical staging system is used to classify patients with HS into three disease severity groups.
  Stage I - abscess formation (single or multiple), no sinus tracts or cicatrization/scarring.
  Stage II - recurrent abscesses with sinus tracts and scarring, single or multiple separated lesions.
  Stage III - diffuse or almost diffuse involvement, or multiple interconnected sinus tracts and abscesses across the entire area
Changes in Dermatology Life Quality Index (DLQI) scores at weeks 4, 8, 12, and 16 compared to baseline. | Baseline, weeks 4, 8, 12, and 16
  A Quality of Life Score will be calculated based upon the Dermatology Life Quality Index (DLQI).
  The DLQI is a validated general dermatology questionnaire that consists of 10 items that assess subject health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). It has been extensively used in dermatology clinical trials for AD. The DLQI is a psychometrically valid and reliable instrument that has been translated into several languages, and the DLQI total scores have been shown to be responsive to change.
  The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Changes in Visual Analogue Scale (VAS) pain scores at weeks 4, 8, 12, and 16 compared to baseline. | Baseline, weeks 4, 8, 12, and 16
  A Pain Score will be calculated based upon a 10-point visual analog pain scale, which has been widely used to rate pain in both children and adults and has also been used in dermatology clinical trials.
  Response based on an improvement from baseline at all scheduled time points will be calculated. We will compare pre and post treatment pain values and categorize patients as (i) Resolved (ii) Improved (iii) Stable (iv) Worsened

OTHER OUTCOMES:
Change from baseline in draining fistula counts at week 16. | Baseline and Week 16
Changes in lesion counts (A, N, AN) at weeks 4, 8, and 12 compared to baseline. | Baseline and weeks 4, 8, and 12
  We will assess the average change in inflammatory lesion count per subject following 4, 8, 12, and 16 weeks of treatment as compared to baseline. Inflammatory lesions are defined as inflammatory nodules or abscesses.
Changes in ulceration at weeks 4, 8, 12, and 16 compared to baseline. | Baseline and weeks 4, 8, 12 and 16
  Secondary exploratory endpoints include change in ulceration and change in overall disease severity by clinical phenotype. No current scoring system exists in HS for ulcerations. Subjects with ulceration present at baseline visit will be assessed for change in ulceration number by anatomical region or size (>25% decrease, >50% decrease, 75% decrease, >90% decrease).
Change in clinical phenotype at week 16 compared to baseline. | Baseline and week 16
  Clinical phenotype of subject (Follicular nodular phenotype vs. infiltrating phenotype vs. comedonal phenotype vs. ulcerating phenotype) will be identified at baseline. Subjects will be reassessed every 4 weeks to identify any shifts in phenotype with therapy. At week 16, descriptive sub- analysis will be performed to identify any clinical phenotypes that are more or less likely to respond to TYK2 inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kimball, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No